CLINICAL TRIAL: NCT03489642
Title: Innovative Pulmonary Rehabilitation Telehealth Program for Improving COPD Patient Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: American Association for Respiratory Care (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00141490
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD Telehealth Program (Experimental): Participants will take part in a structured telehealth program for 12 weeks. Web-based educational tools will be made available to participants. Study participants will meet with a registered respiratory therapist two times per week.
  Interventions: Behavioral: Telehealth Program

INTERVENTIONS:
Behavioral: Telehealth Program — Telehealth program delivered remotely to study participants. Program developed by Cambium Technologies.

SUMMARY:
Researchers want to learn more about telehealth pulmonary rehabilitation programs that help people with Chronic obstructive pulmonary disease (COPD) improve physical activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Hospital discharge diagnosis of COPD
* Spirometry-confirmed evidence of COPD Global Initiative for Chronic Obstructive Lung Disease (GOLD) stages I to IV
* Access to internet connection and knowledge on use of web-based programs

Exclusion Criteria:

* Persons with additional significant comorbidities including cancer, cardiac disease and physical impairments
* Non-English speaking persons
* The inability to provide an informed consent

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Measure of physical activity | Change from Baseline to Week 12
  Changes will be measured using the Yale Physical Activity Survey (YPAS). The tool is composed of two sections - (a) amount of physical activity/exercise performed during a typical week in the past month and (b) activities performed in the past month. The final index score is the sum of five individual indices (vigorous, leisurely walking, moving, standing and sitting). Scores on the scale range from 0 to 137. The higher the score the more active a person.

SECONDARY OUTCOMES:
Quality of Life | Change from Baseline to Week 12
  The COPD Assessment Test (CAT) will be used to measure the health status of the subjects. The test has eight questions. Each question has a range from 0-5. The total score for the test ranges from 0 to 40. The higher the score the more severe a person's COPD.
Adherence to physical activity requirements | Week 12
  Patients receive an individualized exercise plan (minutes and days per week). Adherence to physical activity is assessed by the proportion of weeks subjects achieve their planned physical activity time.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Skinner, RRT, CPFT, Principal Investigator — University of Kansas Medical Center; Dave Burnett, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633